CLINICAL TRIAL: NCT04267523
Title: Effectiveness of a Web-based Intervention on Parental Psychological Flexibility and Emotion Regulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Almeria (Other)
Collaborators: Universitat Jaume I (Other)
Responsible Party: Principal Investigator, Juan Miguel Flujas, Principal Investigator, Universidad de Almeria
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Psy001
Record Dates: First submitted 2019-12-10; First posted 2020-02-13 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Parents
Keywords: Parenting; Psychological flexibility; Third-wave therapies; Web-based intervention; Emotion regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based parenting intervention (Experimental): Families randomized to this intervention group will receive a self-administered web-based parenting intervention. Parents have access to a weekly 6-modules parenting intervention.
  Interventions: Behavioral: Web parenting intervention
- Face-to-face parenting intervention (Active Comparator): Families randomized to this intervention group will receive a face-to-face group parenting intervention. Groups will meet weekly for 120 minutes for 4 weeks.
  Interventions: Behavioral: Group parenting intervention

INTERVENTIONS:
Behavioral: Web parenting intervention — Parents participate in the self-delivered web-based parenting intervention for 6 modules. Treatment includes abilities of psychological flexibility (to be open, aware and active), emotion regulation, and positive parenting strategies.
  Arms: Web-based parenting intervention
Behavioral: Group parenting intervention — Parents participate in face-to-face a weekly 2-hour group for 4 sessions. Treatment includes abilities of psychological flexibility (to be open, aware and active), emotion regulation, and positive parenting strategies.
  Arms: Face-to-face parenting intervention

SUMMARY:
This project aims to validate a web-based clinical intervention for families with children suffering neurodevelopmental or behavioral disorders to promote psychological flexibility and emotion regulation strategies in parents.

DETAILED DESCRIPTION:
Family context, and specifically parents' educational styles (PE) can act as a protective or risk factor for the maintenance and development of various disorders in childhood. When the child is diagnosed of a disease, disorder or difficulty, parents can develop a series of beliefs that will mediate their PEs, their barriers and their emotional repertoire. It can worsen the family climate, lead to maladaptive behaviors, and finally, lead to difficulties in adherence to treatment due to possible avoidance patterns. Several studies indicate that these patterns are mediated by a regulation of dysfunctional emotions in parents by not tolerating the discomfort caused by the suffering of their children.

This project aims to validate a web-based clinical intervention for families with children suffering neurodevelopmental or behavioral disorders to promote psychological flexibility and emotion regulation strategies in parents. Clinical intervention is focused in improving emotion regulation and positive parenting strategies using third-wave/contextual therapies. The intervention consist in 6 sessions with a duration of 1.5 hours. This study compare a a face-to-face parenting intervention group with a web-based parenting intervention. The first hypothesis is that both parental interventions will improve the educational styles, emotional competencies and well-being of parents in pos-test and 3-month follow up assessment. Second, web-based intervention will be more efficient in comparison with face-to-face intervention.

ELIGIBILITY:
Inclusion Criteria:

A. Be a parent/guardian of a child between 0 and 12 years old. B. Be a parent/guardian of a child who obtains a limit score on any of the scales of the Difficulties and Capabilities Questionnaire (SDQ).

C. Obtain a high score in parental inflexibility / emotional distress through the Parental Acceptance Questionnaire in any of its subscales.

D. Parents/guardians have a device that provides access to the web-based intervention.

E. They agree to participate in the study by signing the informed consent

Exclusion Criteria:

A. The parent/guardian is in a process of separation or negligent parenting, this aspect will be assessed from a clinical trial in the initial interview.

B. The parent/guardian has serious psychological or substance use problems or disorders that may hinder their participation in the study.

C. The parent/guardian presents Spanish comprehension barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-05-05 (Estimated)

PRIMARY OUTCOMES:
Parental Acceptance Questionnaire (Flujas-Contreras, García-Palacios, & Gómez, 2018) | Change from baseline at immediately after the intervention, and at 3 months
  To assess Measures psychological flexibility in parents regarding the interaction with their children through 3 dimensions: open, aware and active. Spanish version has internal consistency of .82
Difficulties Emotion Regulation Scale (DERS: Hervás & Jódar, 2008) | Change from baseline at immediately after the intervention, and at 3 months
  To assess the emotional regulation of parents. It consists of 28 items that make up 5 dimensions of emotional deregulation: lack of control, rejection, interference, neglect and confusion. The reliability index (Cronbach's alpha) is between .87 and .93
Parental Stress Scale (PSS; Alonso-Arbiol y Balluerka, 2007) | Change from baseline at immediately after the intervention, and at 3 months
  To assess the level of parental stress. It consists of 20 items that evaluate positive and negative experiences. The scale has a reliability of .77 and .76

SECONDARY OUTCOMES:
Satisfaction with Life Scale (SWLS; Atienza, Pons, Balaguer, & García-Merita, 2000) | Change from baseline at immediately after the intervention months, and at 3 months
  to assess the overall satisfaction of parents as a one-dimensional construct, it consists of 5 items that are answered on a Likert scale of 1 to 7; the Spanish version has provided reliability indexes of .84
Strength and Difficulties Questionnaire, (SDQ; Gómez-Beneyto et al., 2012) | Change from baseline at immediately after the intervention, and at 3 months
  In order to evaluate the effects of the intervention on the behavior of the children, behavioral changes in difficulties, emotional symptoms, behavioral problems, hyperactivity problems, problems with partners and prosocial actions

OTHER OUTCOMES:
Client Satisfaction Questionnaire (Hidalgo y cols., 2013) | Immediately after the intervention
  It consists of 8 items on a 4-point Likert scale that assesses satisfaction in a one-dimensional way
Parental coping and mood | Change from baseline at immediately after the intervention
  The current mood and the perception of coping capacity will be assessed pre and post session through two questions that measure mood by means of visual scale of faces (Likert of 5 points) and coping by Likert scale of 5 points

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Gomez, Prof., Study Director — University de Almeria; Azucena Garcia-Palacios, Prof., Study Director — University Jaume I
Locations (2):
- Spain (2):
  - University of Almería, Almería, Almeria
  - University Jaume I, Castellon, Castellón

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available after deidentification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The duration of the study
Access Criteria: Not decided